CLINICAL TRIAL: NCT00230997
Title: An Open Label 24-Week, Flexible Dose Trial to Assess the Safety and Efficacy of Galantamine in Patients With Dementia With Lewy Bodies
Brief Title: Safety and Efficacy of Galantamine in Patients With Dementia With Lewy Bodies
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Neurological Research Center (Industry)
Collaborators: Ortho-McNeil Neurologics, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GAL-ALZ-421
Record Dates: First submitted 2005-09-29; First posted 2005-10-03 (Estimated); Last update posted 2005-12-16 (Estimated); Status verified 2005-09

CONDITIONS: Lewy Body Disease
Keywords: Galantamine; Dementia with Lewy Bodies; Treatment
MeSH Terms: conditions — Lewy Body Disease | interventions — Galantamine

INTERVENTIONS:
Drug: Galantamine

SUMMARY:
TRIAL SUMMARY:

This is an open-label, 24-week, investigator initiated study to evaluate the safety and efficacy of galantamine (16 8 to 24 mg/day; flexible dosing) in the treatment of Dementia with Lewy bodies. The primary efficacy variables will be the NPI -12, the COGDRAS tests of attention and visuospatial orientation, and the ADCS-CGIC. The secondary efficacy variables will be the MMSE, ADCS-ADL-Inventory, ADAS-Cog, PSQI, and the use of concomitant rescue antipsychotic medication. PET scanning will be obtained on 10 patients at one site. An interim analysis will also be performed. Safety outcome measures will be adverse event reports, vital signs, physical examinations, ECG, laboratory parameters and the UPDRS (motor subscale).

DETAILED DESCRIPTION:
TRIAL DESIGN

1. Rationale

   In a previously published study of DLB treated with rivastigmine, efficacy was seen to be maximized at 20 weeks in multiple parameters compared to placebo. The efficacy was seen in the NPI - 4 as well as the NPI -10, MMSE and a Computerized Cognitive Assessment Systems Score5. There was no change in UPDRS score. The efficacy of rivastigmine for patients with DLB responding greater than 30 percent in behavioral measures was equal to or better than most studies of antipsychotic medications used for behavioral abnormalities in DLB and AD patients.

   Since the titration for galantamine involves less time than the titration for rivastigmine, an interim analysis may show efficacy at 12 weeks. However, for complete efficacy and safety evaluations, a 24-week treatment for galantamine is preferable. Since the cholinergic deficits in DLB patients is more profound than that for AD patients, the dose range of 16 8 to 24 mg/day for DLB patients should be sufficient to show efficacy. Since galantamine has previously been shown to be efficacious in the domains of behavior, cognition, ADL's and global assessment in AD patients, we expect efficacy to be shown similarly and perhaps to a greater extent in DLB patients.

   TREATMENT OF SUBJECTS

   There will be seven visits in this 24-week treatment trial with galantamine for DLB. For all visits a time window of +/- 3 days relative to baseline visit V2 is applicable.

   Screen: Visit 1 (-4 week - 0)

   At visit 1 (V1) subjects will be evaluated for their suitability for enrollment. It is acceptable for this visit to be conducted on more than one day, although it should not be done over longer than a week. Prior to the conduct of any trial related procedures a complete explanation (both verbally and written) of the nature and purpose of the trial will be given by the Investigator (or designee). The subject will be requested to sign and date the IRB/IEC approved Informed Consent. Subject's eligibility for the trial will be determined on the basis of the inclusion/exclusion criteria, and from the results of the following pre-treatment assessments:
   * Medical history
   * Complete neurological examination
   * Complete physical examination
   * CT Scan/MRI
   * Vital signs (blood pressure/heart rate)
   * Weight
   * Height
   * ECG
   * Complete chemistry panel, hematology, B12, folate, RPR, thyroid panels including TSH (if not done within the last 3 months)
   * Urine pregnancy test (if applicable)
   * Concomitant medications
   * Mini Mental State Exam (MMSE)

     * NPI-12
   * PSQI
   * Modified Hachinski Ischemic Scale (MHIS)

   Baseline: Visit 2 (Week 0)

   At the beginning of this visit the Investigator should review all test results from Visit 1, this will include the completion of eligibility criteria. If patient is eligible to continue in the trial, the following assessments will be carried out:

   • Brief physical examination
   * Vital signs (blood pressure/heart rate)
   * Weight
   * Concomitant medications
   * MMSE
   * NPI-12
   * ADAS-Cog
   * ADCS-CGIC
   * FDG-PET*
   * PSQI
   * ADCS-ADL inventory
   * Fluctuation scales
   * UPDRS
   * COGDRAS
   * Dispense medication (See table)
   * AE's

   Titration: Visits 3 (Week 4), Visit 4 (Week 8)

   During the titration visits (Visit 3 and Visit 4) the following assessments will be done:

   • Brief physical examination
   * Vital signs (blood pressure/heart rate) • Weight
   * Concomitant medications
   * NPI-12
   * PSQI
   * Fluctuation scales
   * Dispense medication (See table)
   * AE's
   * Drug accountability

   Maintenance: Visit 5 (Week 12), Visit 6 (Week 20)

   Subjects who have completed the titration phase will continue the 12 week maintenance phase. On clinic visit days subjects will have the following assessments:

   • Brief physical examination

   • Vital signs (blood pressure/heart rate)

   • Weight

   • Concomitant medications

   • MMSE (Visit 5 only)

   • NPI-12

   • ADAS-Cog (Visit 5 only)

   • PSQI

   • ADCS-ADL inventory (Visit 5 only)

   • Fluctuation scales

   • UPDRS (Visit 5 only)

   • COGDRAS (Visit 5 only)

   • Dispense medication (See table)

   • AE's

   • Drug Accountability

   • Efficacy measures (Visit 5 only)

   Final Visit: Visit 7 (Week 24)

   The subject will be scheduled for a clinic visit to perform the final assessments. The following assessments will be carried out:

   • Complete neurological examination

   • Complete physical examination
   * Vital signs (blood pressure/heart rate)
   * Weight
   * ECG
   * Complete chemistry panel and hematology
   * Urine pregnancy test (if applicable)
   * Concomitant medications
   * Mini Mental State Exam (MMSE)
   * NPI-12
   * ADAS-Cog
   * ADCS-CGIC
   * FDG-PET*
   * PSQI
   * ADCS-ADL inventory
   * Fluctuation scales
   * UPDRS
   * COGDRAS
   * Drug accountability

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects (>50 years old) diagnosed with Dementia with Lewy bodies, in accordance with the consensus criteria for probable Dementia with Lewy bodies (McKeith et al., 1996) viii.
* NPI score ≥ 8 at screening
* MMSE ≥ 7 at screening
* Subjects living at home or in a residential or community care home. Subjects who live with or have regular daily visits from a responsible caregiver. Subjects must be able to read, write, and fully understand the language of the scales used in this trial.
* Subjects must exhibit sufficient visual, hearing, and communication capabilities
* The Informed Consent must be given by the subject and the subject's legally acceptable representative.
* The informed consent must also be signed by the caregiver.
* CT or MRI within last 12 months - to be performed if not done

Exclusion Criteria:

* Neurodegenerative disorders such as Alzheimer's disease, Frontotemporal dementia, including Pick's disease, Korsakoff's syndrome, Huntington's chorea, Down's syndrome, Creutzfeldt-Jacob disease and causes of Parkinsonism other than DLB.
* One of the following conditions possibly resulting in cognitive impairment:

  * Acute cerebral trauma, subdural hematoma and injuries secondary to chronic trauma (such as boxing).
  * Hypoxic cerebral damage whether or not due to acute or chronic cerebral hypoperfusion,
  * Vitamin deficiency state such as folate, vitamin B12 and other B complex deficiencies, e.g., thiamine deficiency in Korsakoff's syndrome. Note: subjects taking regular B12 and folate are not necessarily excluded (treatment must be stable, ongoing for at least 4 weeks prior to entry).
  * Infection such as cerebral abscess, neurosyphilis, meningitis or encephalitis.
  * Primary or metastatic cerebral neoplasia.
  * Significant endocrine or metabolic disease e
  * Mental retardation or oligophrenia. Multi-infarct dementia or clinically active cerebrovascular disease
* Subjects with the following co-existing medical condition:

  * Any history of epilepsy or convulsions except for febrile convulsions during childhood.
  * Current clinically significant psychiatric disease, as judged by DSM-IV criteria, in particular current major depression or schizophrenia.
  * Peptic ulcer: if the ulcer is to be considered still "active", i.e., treatment for this condition started <3 months ago or if treatment is not successful (still symptoms present), the subject is not eligible.
  * Clinically significant hepatic, renal, pulmonary, metabolic or endocrine disturbances.
  * Current, clinically significant cardiovascular disease that would be expected to limit the subject's ability to participate in and complete a 7-month trial.
  * Any agent being used for the treatment of dementia (approved, experimental or over the counter agents),
* History of drug or alcohol abuse within the last year or prior prolonged history.
* Female subject of childbearing potential without adequate contraception. Females who are breast-feeding are also excluded.
* Subjects who, in the opinion of the investigator, are otherwise unsuitable for a trial of this type.
* History of severe drug allergy or hypersensitivity; including recorded hypersensitivity to cholinesterase inhibitors, choline agonists or similar agents, bromide or the components of the drug under study.
* Subjects who have previously been enrolled in other galantamine HBr trials. Subjects who were screened for previous galantamine studies but not enrolled may be re-screened for this study.
* Subjects on antipsychotics other than Risperdal® (risperidone), Zyprexa® (olanzapine), Seroquel® (quetiapine), Geodon® (ziprasidone).
* Conditions that could interfere with the absorption of the compound or with the evaluation of the disease.

Min Age: 51 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50
Dates: Start 2002-12; Study Completion 2004-08

PRIMARY OUTCOMES:
NPI-12
ADCS-CGIC
COGDRAS

SECONDARY OUTCOMES:
ADCS-ADL
MMSE
ADAS-Cog
PSQI
Concomitant Antipsychotic Medication use

CONTACTS AND LOCATIONS:
Overall Officials: Keith R Edwards, M.D, Study Director — Neurological Research Center Inc.
Locations (5):
- United States (5):
  - Indiana University for AD and Related Disorders, Indianapolis, Indiana
  - Buffalo Insititute for Medical Research, Buffalo, New York
  - Alzheimer's Center of Pittsburgh, Pittsburgh, Pennsylvania
  - UTHSCSA Psychiatry Department, San Antonio, Texas
  - Neurological Research Center, Inc., Bennington, Vermont

REFERENCES:
- [Background] Tonkopii VD, Prozorovskii VB, Suslova IM. [Interaction of reversible inhibitors with the catalytic centers and allosteric sites of cholinesterases]. Biull Eksp Biol Med. 1976 Aug;82(8):947-50. Russian. PMID 1026294
- [Background] Thomsen T, Kewitz H. Selective inhibition of human acetylcholinesterase by galanthamine in vitro and in vivo. Life Sci. 1990;46(21):1553-8. doi: 10.1016/0024-3205(90)90429-u. PMID 2355800
- [Background] Maelicke A, Albuquerque EX. Allosteric modulation of nicotinic acetylcholine receptors as a treatment strategy for Alzheimer's disease. Eur J Pharmacol. 2000 Mar 30;393(1-3):165-70. doi: 10.1016/s0014-2999(00)00093-5. PMID 10771010
- [Background] Papka M, Rubio A, Schiffer RB. A review of Lewy body disease, an emerging concept of cortical dementia. J Neuropsychiatry Clin Neurosci. 1998 Summer;10(3):267-79. doi: 10.1176/jnp.10.3.267. PMID 9706534
- [Background] Hansen L, Salmon D, Galasko D, Masliah E, Katzman R, DeTeresa R, Thal L, Pay MM, Hofstetter R, Klauber M, et al. The Lewy body variant of Alzheimer's disease: a clinical and pathologic entity. Neurology. 1990 Jan;40(1):1-8. doi: 10.1212/wnl.40.1.1. PMID 2153271
- [Background] Perry RH, Irving D, Blessed G, Fairbairn A, Perry EK. Senile dementia of Lewy body type. A clinically and neuropathologically distinct form of Lewy body dementia in the elderly. J Neurol Sci. 1990 Feb;95(2):119-39. doi: 10.1016/0022-510x(90)90236-g. PMID 2157823
- [Background] Holmes C, Cairns N, Lantos P, Mann A. Validity of current clinical criteria for Alzheimer's disease, vascular dementia and dementia with Lewy bodies. Br J Psychiatry. 1999 Jan;174:45-50. doi: 10.1192/bjp.174.1.45. PMID 10211150
- [Background] McKeith IG, Galasko D, Kosaka K, Perry EK, Dickson DW, Hansen LA, Salmon DP, Lowe J, Mirra SS, Byrne EJ, Lennox G, Quinn NP, Edwardson JA, Ince PG, Bergeron C, Burns A, Miller BL, Lovestone S, Collerton D, Jansen EN, Ballard C, de Vos RA, Wilcock GK, Jellinger KA, Perry RH. Consensus guidelines for the clinical and pathologic diagnosis of dementia with Lewy bodies (DLB): report of the consortium on DLB international workshop. Neurology. 1996 Nov;47(5):1113-24. doi: 10.1212/wnl.47.5.1113. PMID 8909416
- [Background] McKeith IG, Ballard CG, Perry RH, Ince PG, O'Brien JT, Neill D, Lowery K, Jaros E, Barber R, Thompson P, Swann A, Fairbairn AF, Perry EK. Prospective validation of consensus criteria for the diagnosis of dementia with Lewy bodies. Neurology. 2000 Mar 14;54(5):1050-8. doi: 10.1212/wnl.54.5.1050. PMID 10720273
- [Background] Perry EK, Marshall E, Perry RH, Irving D, Smith CJ, Blessed G, Fairbairn AF. Cholinergic and dopaminergic activities in senile dementia of Lewy body type. Alzheimer Dis Assoc Disord. 1990 Summer;4(2):87-95. PMID 2357341
- [Background] Perry EK, Irving D, Kerwin JM, McKeith IG, Thompson P, Collerton D, Fairbairn AF, Ince PG, Morris CM, Cheng AV, et al. Cholinergic transmitter and neurotrophic activities in Lewy body dementia: similarity to Parkinson's and distinction from Alzheimer disease. Alzheimer Dis Assoc Disord. 1993 Summer;7(2):69-79. doi: 10.1097/00002093-199307020-00002. PMID 8347330
- [Background] Shiozaki K, Iseki E, Uchiyama H, Watanabe Y, Haga T, Kameyama K, Ikeda T, Yamamoto T, Kosaka K. Alterations of muscarinic acetylcholine receptor subtypes in diffuse lewy body disease: relation to Alzheimer's disease. J Neurol Neurosurg Psychiatry. 1999 Aug;67(2):209-13. doi: 10.1136/jnnp.67.2.209. PMID 10406992
- [Background] McKeith IG, Grace JB, Walker Z, Byrne EJ, Wilkinson D, Stevens T, Perry EK. Rivastigmine in the treatment of dementia with Lewy bodies: preliminary findings from an open trial. Int J Geriatr Psychiatry. 2000 May;15(5):387-92. doi: 10.1002/(sici)1099-1166(200005)15:53.0.co;2-9. PMID 10822236
- [Background] McKeith I, Del Ser T, Spano P, Emre M, Wesnes K, Anand R, Cicin-Sain A, Ferrara R, Spiegel R. Efficacy of rivastigmine in dementia with Lewy bodies: a randomised, double-blind, placebo-controlled international study. Lancet. 2000 Dec 16;356(9247):2031-6. doi: 10.1016/S0140-6736(00)03399-7. PMID 11145488
- [Background] Shea C, MacKnight C, Rockwood K. Donepezil for treatment of dementia with Lewy bodies: a case series of nine patients. Int Psychogeriatr. 1998 Sep;10(3):229-38. doi: 10.1017/s1041610298005341. PMID 9785144
- [Background] Cummings JL. Cholinesterase inhibitors: A new class of psychotropic compounds. Am J Psychiatry. 2000 Jan;157(1):4-15. doi: 10.1176/ajp.157.1.4. PMID 10618007
- [Result] Edwards KR, Hershey L, Wray L, Bednarczyk EM, Lichter D, Farlow M, Johnson S. Efficacy and safety of galantamine in patients with dementia with Lewy bodies: a 12-week interim analysis. Dement Geriatr Cogn Disord. 2004;17 Suppl 1:40-8. doi: 10.1159/000074681. PMID 14676468
- [Result] Edwards K, Farlow M, Hake A et al. An Open Label 24-Week, Flexible Dose Trial to Assess the Safety and Efficacy of Galantamine in Patients with Dementia with Lewy Bodies. Neurobiology of Aging. 2004; 25 (S2): 21.
- [Result] Edwards K, Hershey L, Farlow M, Lichter D, Johnson S: Galantamine for the treatment of dementia with Lewy bodies. Movement Disorders: S336, Vol 19/Suppl 9, 2004